CLINICAL TRIAL: NCT06123715
Title: PeRiOperative VItamin C to Reduce perSistent paIn After tOtal kNee Arthroplasty (PROVISION): a Pilot Multicentre Randomized Controlled Trial
Brief Title: Perioperative Vitamin C to Reduce Persistent Pain After Total Knee Arthroplasty
Acronym: PROVISION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Arthritis Society, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-5642
Record Dates: First submitted 2023-10-10; First posted 2023-11-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Knee Pain Chronic; Post Operative Pain
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative | interventions — Ascorbic Acid; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Preoperative Vitamin C capsules
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): Preoperative placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — Drug: Patients in the intervention group will receive 2g Vitamin C orally within 4 hours of the start of the surgery followed by 500 mg of Vitamin C to be taken orally twice a day from post-op day1 to day 56.
  Other Names: Ascorbic Acid
  Arms: Intervention
Drug: Placebo — Drug: Patients in the placebo group will receive identical placebo capsules taken orally within 4 hours of the start of the surgery followed by placebo capsules taken orally twice a day from post-op day 1 to day 56.
  Other Names: Lactose (Monohydrate)
  Arms: Placebo

SUMMARY:
Phase II Multicentre, pilot, parallel-group, blinded, 1:1 randomized controlled trial to determine the feasibility of conducting a larger definitive trail of using vitamin C to reduce persistent pain in patients undergoing total knee arthroplasty surgery.

DETAILED DESCRIPTION:
PROVISION is a multicentre, pilot, parallel-group, blinded, randomized controlled trial of 300 patients undergoing total knee arthroplasty surgery. Consented eligible patients will be randomized to receive vitamin C: 2000 mg taken orally within 4 hours of the start of surgery, followed by 500 mg of vitamin C taken twice daily from post-operative day 1 to day 56 (8 weeks). Patient in the control group will receive placebo lactose monohydrate capsules. Study medications will be prepared to look similar and labelled as per regulatory requirements. Patients will follow up on post-operative days 1-3, weeks 2,4,6, and 8 post-operatively, and at 3- and 12-months post-operatively to report on pain, opioid and analgesic consumption, medication adherence, adverse events, functional, mood, and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Undergoing a unilateral or bilateral primary total knee arthroplasty for advanced osteoarthritis of the knee

Exclusion Criteria:

* TKA for infection (septic joint), fracture, ankylosing spondylitis, lupus, or psoriatic arthritis
* History of kidney stones, acute or chronic renal failure, hemochromatosis, or glucose-6-phosphate deficiency
* Unlikely to comply with follow-up (e.g., no fixed address, plans to move out of town)
* Language difficulties that would impede valid completion of questionnaires
* Planned staged bilateral TKA
* Treating surgeon deems patient inappropriate for inclusion in trial
* Any allergy or sensitivity to milk
* Pregnant or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Study will determine feasibility of enrolling, recruiting, and follow-up with patients. | 12 months
  The study will assess the feasibility of enrolling, recruiting, and following-up with patients undergoing a primary total knee arthroplasty (TKA) through active monitoring of recruitment/enrollment rates on a monthly basis for a total of one year using excel trackers. The follow-up rate of patients will be assessed at 12 months based on completion of all 12 month questionnaires.
Clinical site compliance | 12 months
  Clinical site compliance with trial protocol will be determined based on number of protocol deviations at each site as logged on the deviation logs. This will be assessed on a monthly basis for a full year to maintain active monitoring of compliance.
Resource Assessment | 12 months
  This pilot study will help determine the resources required for larger definitive trial based on critical analysis of recruitment trackers to assess time spent on recruitment/enrollment.

SECONDARY OUTCOMES:
Prevalence of persistent pain | 3 months and 12 months
  Pain intensity measured using 0-10 Numeric Rating Scale (NRS) scale at rest and movement
Qualities and characteristics of persistent pain | 3 months and 12 months
  Pain qualities measured using the 0-10 scale of the Short Form McGill Pain Questionnaire 2 (SF-MPQ-2)
Persistent Neuropathic Pain | 3 months and 12 months
  Neuropathic pain assessed on a binary scale of Yes or No using the Douleur Neuropathique 4 (DN4) symptoms interview
Acute and chronic analgesic consumption | Day of surgery, post-operative day 1-3, 3 months, and 12 months
  Analgesic and oral morphine-equivalent opioid consumption
Development of Complex Regional Pain Syndrome (CRPS) | 3 months and 12 months
  Presence of CRPS measured by a physical assessment of sensory, vasomotor, sudomotor/edema, and motor/tropic categories using the Budapest Criteria
Physical function | 3 months and 12 months
  Patient reported outcome measure to assess level of function, daily living activities and their affect on pain measured by answering 12 questions using the Oxford Knee Score (OKS)
Emotional functioning | 3 months and 12 months
  Patients emotional functioning measured on a scale of 1-5 using the EQ-5D-5L
Patient Satisfaction | 3 months and 12 months
  Assessment of patient satisfaction with surgery on scale of 0-100
Quality of life assessment | 3 months and 12 months
  Patient reported assessment of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a scale of level 1 - level 5 using the EuroQol 5-dimension 5-level (EQ-5D-5L)
Adverse events | 3 months and 12 months
  Monitored as a secondary safety outcome using an assessment of follow-up visits for drug related adverse events and passive surveillance of clinical notes

CONTACTS AND LOCATIONS:
Overall Officials: James Khan, MD, Principal Investigator — University Health Network; Department of Anesthesia and Pain Medicine; Raman Mundi, MD, Principal Investigator — Holland Orthopedic and Arthritic Centre; Harman Chaudhry, MD, Principal Investigator — Holland Orthopedic and Arthritic Centre; Jesse Wolfstadt, MD, Principal Investigator — Mount Sinai Hospital; Department of Surgery
Locations (3):
- Canada (3):
  - Sunnybrook - Holland Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No